CLINICAL TRIAL: NCT04395365
Title: Primary Antibiotic Prophylaxis Using Co-trimoxazole to Prevent Spontaneous Bacterial Peritonitis in Cirrhosis
Acronym: ASEPTIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17/0894
Record Dates: First submitted 2020-04-18; First posted 2020-05-20 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Co-trimoxazole (Experimental): Co-trimoxazole, 960mg capsule oral tablet, to be taken daily for 18 months
  Interventions: Drug: Co-Trimoxazole 960Mg Dispersible Tablet
- Placebo (Placebo Comparator): Placebo, 960mg capsule oral tablet, to be taken daily for 18 months
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Co-Trimoxazole 960Mg Dispersible Tablet — Antibiotic prophylaxis of Spontaneous Bacterial Peritonitis
  Arms: Co-trimoxazole
Drug: Placebo oral tablet — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
A multicentre, interventional, double-blind, placebo-controlled, parallel-arm, phase 3, randomised controlled trial to evaluate the use of co-trimoxazole as primary prophylaxis for spontaneous bacterial peritonitis to improve overall survival

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion criteria:

1. Patients with Child-Pugh Class B or C cirrhosis and presence of ascites requiring any diuretic treatment or at least 1 or more paracentesis within 3 months prior to enrolment.
2. Patient at least 18 years of age
3. Documented informed consent to participate

Exclusion criteria:

1. Patients with current or previous Spontaneous Bacterial Peritonitis (defined as ascitic polymorphonuclear (PMN) cell count >250/mm3 with either positive or negative ascitic fluid culture without evident intra-abdominal surgically treatable source of infection. A white cell count >500 cell/mm2 or positive microbial culture may be considered as evidence of previous SBP if the site PI considers this was in the context of a likely clinical diagnosis of SBP).
2. Patients receiving palliative care with an expected life expectancy of <8 weeks
3. Allergic to co-trimoxazole, trimethoprim or sulphonamides
4. Pregnant or lactating mothers
5. Patient enrolled in a clinical trial of investigational medicinal products (IMPs) that would impact on their participation in the study
6. Patients with serum potassium (>5.5 mmol/L) related to pre-existing kidney disease which cannot be reduced*
7. Patients receiving antibiotic prophylaxis (except for rifaximin)*
8. Patients with long-term ascites drains*
9. Women of child-bearing potential and males with a partner of child-bearing potential without effective contraception for the duration of trial treatment
10. Patients with pathological blood count changes

    1. Patients with haemoglobin (Hb) <70g/L*
    2. Granulocytopenia defined as absolute neutrophil counts of less than 500 cells per microliter*
    3. Severe thrombocytopenia with a platelet count <30 x109 /L*
11. Patients with severe renal impairment, with eGFR <15 ml/min*
12. Patients with skin conditions: exudative erythema multiform, Stevens-Johnson syndrome, toxic epidermal necrolysis and drug eruption with eosinophilia and systemic symptoms
13. Patients with congenital conditions: congenital glucose-6-Phosphate dehydrogenase deficiency of the erythrocytes, haemoglobin anomalies such as Hb Köln and Hb Zürich
14. Patients with acute porphyria
15. Any clinical condition which the investigator considers would make the patient unsuitable for the trial.

    * It is common for these investigations to change in patients with cirrhosis and long-term ascitic drains may be removed. Patients can be re-screened for eligibility if this occurs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | The maximum possible period of follow up will be 48 months (assuming a recruitment period of 30 months and 18 months treatment period for final patient recruited)
  Overall Survival

SECONDARY OUTCOMES:
Spontaneous Bacterial peritonitis | Minimum period of 18 months from randomisation
  Time to first incidence of spontaneous bacterial peritonitis (SBP)
Hospital admissions | Minimum period of 18 months from randomisation
  Hospital admission rates
C. difficile-associated diarrhoea | Minimum period of 18 months from randomisation
  Incidence of C. difficile-associated diarrhoea
Infections other than spontaneous bacterial peritonitis with hospital admission | Minimum period of 18 months from randomisation
  Incidence of infections other than spontaneous bacterial peritonitis with hospital admission.
Cirrhosis related events | Minimum period of 18 months from randomisation
  Incidence of other cirrhosis related events (e.g. variceal haemorrhage)
Renal dysfunction | Minimum period of 18 months from randomisation
  Incidence of renal dysfunction with creatinine >133 μmol/L (1.5mg/dL) at any point during hospital admission
Anti-microbial resistance | Minimum period of 18 months from randomisation
  Incidence of anti-microbial resistance
Liver transplantation | Minimum period of 18 months from randomisation
  Incidence of liver transplantation
Liver disease assessed by increase in MELD score | Minimum period of 18 months from randomisation
  Progression of liver disease assessed by increase in MELD score between baseline and end of trial follow up.
Safety and treatment-related serious adverse events | Minimum period of 18 months from randomisation
  Safety and treatment-related serious adverse events
Treatment adherence | Minimum period of 18 months from randomisation
  Treatment adherence (assessed by MARS questionnaire)
Health-related quality of life | Minimum period of 18 months from randomisation
  Health-related quality of life assessed using EQ-5D-5L questionnaire
Health and social care | Minimum period of 18 months from randomisation
  Health and social care resource use assessed using Hospital Episode Statistics (HES) database
Mean incremental cost per quality adjusted life year gained (QALY) | Minimum period of 18 months from randomisation
  Mean incremental cost per quality adjusted life year gained (QALY)
Incidence of resolution of ascites with diuretic treatment not required for 6 months | Minimum period of 18 months from randomisation
  Incidence of resolution of ascites with diuretic treatment not required for 6 months
Transjugular intrahepatic portosystemic shunt (TIPS) insertion | Minimum period of 18 months from randomisation
  Incidence of Transjugular intrahepatic portosystemic shunt (TIPS) insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free hospital, Hampstead, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No